CLINICAL TRIAL: NCT03631394
Title: The Effects of Dietary Nitric Oxide and Anthocyanins on Anaerobic Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Edward Bitok, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5180190
Record Dates: First submitted 2018-06-19; First posted 2018-08-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beetroot and anthocyanin (Experimental): A compound pharmacy will formulate capsules with nitrates extracted from beetroot and anthocyanins from tart cherries. A daily dose of the capsules will be taken for 7 days after the washout period. Each dose will comprise 500 mg of nitrates and 450 mg of anthocyanins. In a meta-review by Dominguez and colleagues, 6-8 mmol of nitrates from beetroot was associated with increased exercise performance. Another review by Kelley et al., showed that marathon runners and resistance trainers ingesting between 450-480 mg of anthocyanins had reduced muscle soreness and decreased oxidative stress. Subject will consume each supplement orally with only water 2 hours pre-prandial.
  Interventions: Other: beetroot and anthocyanin
- beetroot and placebo (Placebo Comparator): The same compound pharmacy will formulate capsules with nitrate extracted from beetroot and a placebo element made of starch. This product will taste the same as the nitrate and anthocyanin supplementation. A daily dose of the capsules will be taken for 7 days after the washout period. Each supplementation will have 500 mg of nitrate and 450 mg of placebo. Subjects will consume each supplement orally with only water 2 hours pre-prandial.
  Interventions: Other: beetroot and placebo

INTERVENTIONS:
Other: beetroot and anthocyanin — Beetroot and anthocyanin will be taken for 7 days during the study two hours prior to eating.
  Arms: beetroot and anthocyanin
Other: beetroot and placebo — Beetroot and placebo will be taken for 7 days during the study two hours prior to eating.
  Arms: beetroot and placebo

SUMMARY:
The purpose of this graduate student research study is to investigate the effects of nitrate from beetroot powder with additional anthocyanins from tart cherry on exercise performance in healthy Loma Linda University students utilizing the Wingate Anaerobic test on stationary bike.

DETAILED DESCRIPTION:
A randomized controlled double-blind crossover study with a baseline and two interventions. On day 1 (baseline), all subjects will have a lactate fingerstick measurement before and after the Wingate protocol. A random subsample (1/3 of subjects) will have 10 milliliters (2 teaspoon) of blood drawn for determination of serum allantoin. Subjects will then be equipped with a pulse oximeter and a heart rate monitor after which they will perform the Wingate Anaerobic test protocol. The protocol includes: 4 minutes of warm up, 3 seconds of warm up sprint with weights, 1-minute relaxed cycling, 2-minute rest, then 10 seconds cycling without weights. This will be followed by 30 seconds sprint with weights and end with 2 minutes of relaxed cycling. A post-activity blood draw will be performed for another 10 milliliters (2 teaspoon) of blood from the same one-third of subjects previously sampled. After baseline data collection, subjects will undergo a 1-week washout (avoiding high antioxidant foods) after which they will be randomized to treatment groups. On day 9, subjects will begin supplementation with nitrate from beetroot powder with additional anthocyanins, or nitrate from beetroot powder with a placebo for 7 days. On day 15 the subject will again repeat the same procedures as day 1, followed by another week of washout. They will supplement again on day 23 and repeat the same procedure as the first intervention on day 29.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Loma Linda University students aged between 21 and 35 years old
* Willing to abstain from caffeine, mouthwash, chewing gums, and high antioxidant foods during the week of supplementation.

Exclusion Criteria:

* Diabetic
* having salivary gland disorder, cardiovascular disease or orthopedic injuries
* pregnant or breastfeeding
* taking NSAIDS
* have an allergy to anthocyanins and/or beetroot
* women who are on their menses

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in blood lactate levels | Day 1
  Participants in this study should reach an anaerobic state as they perform the Wingate test. This lactate pro analyzer will be a tool to examine the participant's change in blood lactate levels by means of POC fingertip lactate measurement. Lactate levels will be measured in all participants at baseline, before and after Wingate Anaerobic test.
Change in blood lactate levels | Day 15
  Participants in this study should reach an anaerobic state as they perform the Wingate test. This lactate pro analyzer will be a tool to examine participant's change in blood lactate levels by means of POC fingertip lactate measurement. Lactate levels will be measured in all participants at intervention I, before and after Wingate Anaerobic test.
Change in blood lactate levels | Day 29
  Participants in this study should reach an anaerobic state as they perform the Wingate test. This lactate pro analyzer will be a tool to examine participant's change in blood lactate levels by means of POC fingertip lactate measurement. Lactate levels will be measured in all participants at intervention II, before and after Wingate Anaerobic test.

SECONDARY OUTCOMES:
Allantoin blood level | Baseline, day 15, and day 29
  Non-fasting blood tests will be done for allantoin during baseline, intervention I, and intervention II.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bitok, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States